CLINICAL TRIAL: NCT04780581
Title: MP3-pulses-COVID-19. Methylprednisolone Pulses Versus Dexamethasone According RECOVERY Protocol in Patients With Pneumonia Due to SARS-COV-2 Coronavirus Infection
Brief Title: Glucocorticoid Therapy in Coronavirus Disease COVID-19 Patients
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Impossibility of reaching the sample size established by protocol
Sponsor: Fundación Instituto de Estudios de Ciencias de la Salud de Castilla y León (Other)
Collaborators: Instituto de Investigación Biomédica de Salamanca (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MP3-pulses-COVID-19; 2020-005026-28 (EudraCT Number)
Record Dates: First submitted 2021-02-15; First posted 2021-03-03 (Actual); Results first posted 2025-01-06 (Actual); Last update posted 2025-01-06 (Actual); Status verified 2024-12

CONDITIONS: Corona Virus Infection
MeSH Terms: conditions — Coronavirus Infections | interventions — Dexamethasone; Salvage Therapy; Methylprednisolone; NOP-bolus regimen

STUDY DESIGN:
Intervention Model Description: Open-label, randomised clinical trial comparing 2 active treatments. Low-intervention clinical trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RECOVERY (Active Comparator): intermediate-dose dexamethasone (6mg/24h - 10 days)
  Interventions: Drug: Dexamethasone
- BOLUS (Experimental): high-dose methylprednisolone bolus (250mg/4h - 3 days)
  Interventions: Drug: Methylprednisolone

INTERVENTIONS:
Drug: Dexamethasone — 6 mg/24h - 10 days
  Other Names: Recovery
  Arms: RECOVERY
Drug: Methylprednisolone — 250 mg/ 24h - 3 days
  Other Names: Bolus
  Arms: BOLUS

SUMMARY:
Treatment with glucocorticoids in COVID patients. Low-intervention, phase IV, open-label, randomised, low-intervention clinical trial comparing 2 active treatments.

DETAILED DESCRIPTION:
The use of high-dose bolus glucocorticoids in the treatment of patients with COVID-19 infection will increase the anti-inflammatory effect without increasing side effects. This will allow a better patient outcome, reducing the number of deaths and the need for intubation or admission to the Intensive Care Unit.

ELIGIBILITY:
Inclusion Criteria:

1. Over 18 years of age
2. Inpatient
3. Diagnosis of SARS-CoV-2 infection confirmed by reverse transcriptase polymerase chain reaction (RT-PCR) or antigen
4. They present evidence in computerized axial tomography (CT) of pulmonary involvement attributed to the infection by COVID. Patients in whom CT scans are not performed must have suspected pulmonary involvement by clinical examination with simple compatible or suggestive radiology.
5. Requires supplementary oxygen due to basal saturation ≤ 93% (with ambient O2, 21%)

Exclusion Criteria:

1. The patient's situation is so serious that the doctor in charge thinks he could die within 24 hours.
2. At the time of randomisation, patients require one of the following 4 ventilatory supports:

   1. high-flow oxygen devices.
   2. non-invasive mechanical ventilation.
   3. invasive mechanical ventilation.
   4. Extracorporeal membrane oxygenation (ECMO).
3. The patient is or has been treated in the 2 weeks prior to randomisation with glucocorticoids or inflammation modifying drugs, both conventional (thiopurines, cyclophosphamide, cyclosporine, tacrolimus), leflunomide, methotrexate, mycophenolate mofetil/mycophenolic acid, sulfasalazine, hydroxychloroquine or chloroquine) as synthetics or biologics directed against therapeutic targets (abatacept, belimumab, CD-20, IL1, IL6, Il12. 23, IL-23, Il.17, TNF, integrin α4β7 or Janus kinase inhibitors JAK). Patients who are only on maintenance treatment with doses of steroids less than or equal to 7.5 mg of prednisone or equivalent per day will not be excluded.
4. The patient is pregnant or breastfeeding.
5. The patient has a chronic renal disease is stage 4 or 5 (CCr <30 ml/min).
6. Moderate to severe dementia at the investigator's discretion.
7. Hypersensitivity to any of the active ingredients or to any of the excipients included in its formulation.
8. Untreated systemic infections not caused by COVID-19.
9. Active stomach or duodenal ulcer.
10. Recent vaccination with live vaccines.
11. Other infection or disease that explains the lung disorder.
12. Inability of the patient to understand the study or to sign the informed consent unless consent is delegated to a legal representative.
13. Active participation in another clinical study in the last 15 days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2021-11-09 (Actual); Study Completion 2021-11-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Luis Corral Gudino, Principal Investigator — Investigator
Locations (4):
- Spain (4):
  - Complejo Asistencial Universitario de León, León
  - Complejo Asistencial Universitario de Salamanca, Salamanca
  - Hospital Clínico Universitario de Valladolid, Valladolid
  - Hospital Universitario Río Hortega, Valladolid

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The sample size estimation (295 patients) for the primary outcomes was based on data from the first waves of COVID-19. Changes in pandemia status triggered to our initial estimation for sample size calculation was outdated. In addition to the high percentage of people vaccinated in Spain, in the summer of 2021 was the end of the fifth wave of COVID-19, with a very small number of patients hospitalized, so the clinical trial was premature ended in August 2021.
Pre-assignment Details: Randomisation was performed using a centralised, computer-generated allocation, stratified by trial site and by age under 70 years, in a 1:1 ratio. 158 patients were assessed for eligibility, and 128 were randomised: 64 to BOLUS group and 64 to RECOVERY group.
Groups:
- BOLUS: high-dose methylprednisolone bolus (250mg/24h - 3 days)
  Methylprednisolone: 250 mg/ 24h - 3 days
Period: Full Modified Intention-to-treat Anal.
Arm/Group | BOLUS | RECOVERY
Started | 64 | 64
Completed | 63 | 62
Not Completed | 1 | 2
Not completed — Protocol Violation | 1 | 2
Period: Follow up to 28 Days (Primary End Point)
Arm/Group | BOLUS | RECOVERY
Started | 63 | 62
Completed | 63 | 62
Not Completed | 0 | 0
Period: Overall Study (90 Days)
Arm/Group | BOLUS | RECOVERY
Started | 63 | 62
Completed (Follow up completed at 90 days) | 63 | 60
Not Completed | 0 | 2
Not completed — Lost to Follow-up | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- BOLUS: high-dose methylprednisolone bolus (250mg/24h - 3 days)
  Methylprednisolone: 250 mg/24h - 3 days
- Total: Total of all reporting groups
Arm/Group | BOLUS | RECOVERY | Total
Number analyzed (Participants) | 63 | 62 | 125
Age, Customized [Count of Participants; unit: Participants]
  18-69 years | 40 | 42 | 82
  70 years and over | 23 | 20 | 43
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 21 | 41
  Male | 43 | 41 | 84
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Hypertension [Count of Participants; unit: Participants] | 31 | 22 | 53
Diabetes [Count of Participants; unit: Participants] | 13 | 10 | 23
Dyslipidaemia [Count of Participants; unit: Participants] | 16 | 22 | 38
COVID-19 characteristics [Count of Participants; unit: Participants]
  Fever | 47 | 43 | 90
  Arthralgia/Myalgia | 21 | 19 | 40
  Cough | 47 | 43 | 90
  Thoracic pain | 8 | 7 | 15
  Nausea | 13 | 10 | 23
  Diarrhoea | 18 | 16 | 34
  Hyposmia/hypogeusia | 10 | 13 | 23
  Headache | 15 | 9 | 24

OUTCOME MEASURES:

1. Primary Outcome: Mortality Rate
Description: Mortality rate (percentage) in COVID-19 patients after high-dose methylprednisolone bolus administration versus mortality rate intermediate-dose dexamethasone pattern (RECOVERY trial)
Time Frame: 28 days
Population: This outcome, mortality rate, was evaluated 28 days after treatment (63 participants in bolus arm vs. 62 participants in recovery arm).
Measure: Count of Participants; unit: Participants
Arm/Group | BOLUS | RECOVERY
Number analyzed (Participants) | 63 | 62
Participants | 3 | 3
Statistical Analysis 1: Comparison: BOLUS vs RECOVERY; Null hypothesis of equal survival curves. Estimates of rate and risk ratios are shown with 95% confidence intervals. All the p-values are 2-sided and shown without adjustment for multiple testing, and p < 0.05 was considered statistically significant. The analyses were performed using IBM SPSS Statistics for Windows, Version 26.0 (Armonk, NY, USA: IBM Corp.); Test type: Equivalence — log-rank statistic test; p = 0.984, Log Rank; Odds Ratio (OR) = 1.0, 95% CI 2-sided [0.2 to 5.1]
Statistical Analysis 2: Comparison: BOLUS vs RECOVERY; Test type: Equivalence — Log-rank method; Risk Difference (RD) = 0.1, 95% CI 2-sided [-8.8 to 9.1]

2. Secondary Outcome: Admission in Intensive Unit Care (ICU)
Description: Number of patients who have been admitted to the ICU.
Time Frame: 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | BOLUS | RECOVERY
Number analyzed (Participants) | 63 | 62
Participants | 10 | 9
Statistical Analysis 1: Comparison: BOLUS vs RECOVERY; Test type: Equivalence — Cochran-Mantel-Haenszel test; p = 0.833, Chi-squared; Odds Ratio (OR) = 1.1, 95% CI 2-sided [0.4 to 3.0]
Statistical Analysis 2: Comparison: BOLUS vs RECOVERY; Test type: Equivalence — Cochran-Mantel-Haenszel test; Risk Difference (RD) = -1.4, 95% CI 2-sided [-14.2 to 11.5]

3. Secondary Outcome: Evaluation of Respiratory Support Requirements
Description: * Proportion of patients (number of cases with respiratory support requirement / total number of patients) with non-invasive mechanical ventilation and/or high-flow oxygen requirements.
  * Proportion of patients (number of cases with respiratory support requirement / total number of patients) with invasive mechanical ventilation or intubation requirements.
Time Frame: 28 days
Measure: Number; unit: proportion of participants
Arm/Group | BOLUS | RECOVERY
Number analyzed (Participants) | 63 | 62
proportion of participants
  invasive mechanical ventilation or intubation requirements | 0.13 | 0.12
  non-invasive mechanical ventilation | 0.05 | 0.03
  high-flow oxygen requirements. | 0.10 | 0.13
Statistical Analysis 1: Comparison: BOLUS vs RECOVERY; non-invasive mechanical ventilation; Test type: Equivalence — Cochran-Mantel-Haenszel test; p = 0.661, Chi-squared; Odds Ratio (OR) = 1.5, 95% CI 2-sided [0.2 to 9.3]
Statistical Analysis 2: Comparison: BOLUS vs RECOVERY; non-invasive mechanical ventilation; Test type: Equivalence — Cochran-Mantel-Haenszel test; Risk Difference (RD) = 1.5, 95% CI 2-sided [-10.2 to 6.9]
Statistical Analysis 3: Comparison: BOLUS vs RECOVERY; high-flow oxygen requirements; Test type: Equivalence — Cochran-Mantel-Haenszel test; p = 0.549, Chi-squared; Odds Ratio (OR) = 0.7, 95% CI 2-sided [0.2 to 2.2]
Statistical Analysis 4: Comparison: BOLUS vs RECOVERY; high-flow oxygen requirements; Test type: Equivalence — Cochran-Mantel-Haenszel test; Risk Difference (RD) = 3.4, 95% CI 2-sided [-8.2 to 15.1]
Statistical Analysis 5: Comparison: BOLUS vs RECOVERY; Invasive mechanical ventilation or intubation requirements analysis; Test type: Equivalence — Cochran-Mantel-Haenszel test; p = 0.809, Chi-squared; Odds Ratio (OR) = 1.1, 95% CI 2-sided [0.4 to 3.3]
Statistical Analysis 6: Comparison: BOLUS vs RECOVERY; Invasive mechanical ventilation or intubation requirements analysis; Test type: Equivalence — Cochran-Mantel-Haenszel test; Risk Difference (RD) = -1.0, 95% CI 2-sided [-13.0 to 11.1]

4. Secondary Outcome: Days in Hospital
Description: Number of days in hospital from the star of the treatment until discharge
Time Frame: 28 days
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | BOLUS | RECOVERY
Number analyzed (Participants) | 63 | 62
Days | 13 (16) | 13 (12)
Statistical Analysis 1: Comparison: BOLUS vs RECOVERY; Test type: Equivalence — T-test; p = 0.908, t-test, 1 sided; Risk Difference (RD) = -0.3, 95% CI 2-sided [-5 to 5]

5. Secondary Outcome: Evaluation of Presence of Adverse Events Related With Use of High Dose of Glucocorticoids.
Description: Occurrence of infections, hyperglycaemia, psychotic states or other adverse effects, if applicable
Time Frame: 28 days
Population: This adverse events related with use of high dose of glucocorticoids and were evaluated 28 days after treatment (63 participants in bolus arm vs. 62 participants in recovery arm).
Measure: Number; unit: Events
Units Other Than Participants: Events
Arm/Group | BOLUS | RECOVERY
Number analyzed (Participants) | 63 | 62
Number analyzed (Events) | 102 | 51
Events
  Secondary infections | 7 | 8
  Hyperglycaemia | 17 | 5
  Psychotic states | 1 | 0
  Other adverse effects no related with use of high dose of glucocorticoids. | 77 | 38
Statistical Analysis 1: Comparison: BOLUS vs RECOVERY; Secondary infections; Test type: Equivalence — Cochran-Mantel-Haenszel test; p = 0.758, Chi-squared; Odds Ratio (OR) = 0.8, 95% CI 2-sided [0.3 to 2.5]
Statistical Analysis 2: Comparison: BOLUS vs RECOVERY; Secondary infections; Test type: Equivalence — Cochran-Mantel-Haenszel test; Risk Difference (RD) = 1.8, 95% CI 2-sided [-10.1 to 13.7]
Statistical Analysis 3: Comparison: BOLUS vs RECOVERY; Hyperglycaemia; Test type: Equivalence — Cochran-Mantel-Haenszel test; p = 0.007, Chi-squared; Odds Ratio (OR) = 4.2, 95% CI 2-sided [1.4 to 12.3]
Statistical Analysis 4: Comparison: BOLUS vs RECOVERY; Hyperglycaemia; Test type: Equivalence — Cochran-Mantel-Haenszel test; Risk Difference (RD) = -18.9, 95% CI 2-sided [-31.8 to -5.6]
Statistical Analysis 5: Comparison: BOLUS vs RECOVERY; Psychotic states; Test type: Equivalence — Cochran-Mantel-Haenszel test; p = 0.319, Chi-squared; Risk Difference (RD) = -1.6, 95% CI 2-sided [-8.5 to 4.4]

6. Secondary Outcome: Evaluation of Other Immunosuppressors Requirements.
Description: Occurrence of use of other immunosuppressors, if applicable
Time Frame: 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | BOLUS | RECOVERY
Number analyzed (Participants) | 63 | 62
Participants | 14 | 14
Statistical Analysis 1: Comparison: BOLUS vs RECOVERY; Test type: Equivalence — Cochran-Mantel-Haenszel test; p = 0.962, Chi-squared; Odds Ratio (OR) = 1.0, 95% CI 2-sided [0.4 to 2.3]
Statistical Analysis 2: Comparison: BOLUS vs RECOVERY; Test type: Equivalence — Cochran-Mantel-Haenszel test; Risk Difference (RD) = 0.4, 95% CI 2-sided [-14.2 to 14.9]

7. Secondary Outcome: Status According to the World Health Organization (WHO) 10-category Scale.
Description: Clinical evaluation of patient status according to the WHO 10-category scale. Minimum value: 1 and maximum value: 10, higher scores mean a worse outcome.
Time Frame: 90 days
Measure: Number; unit: participants
Arm/Group | BOLUS | RECOVERY
Number analyzed (Participants) | 63 | 60
participants
  Dead (10) | 6 | 4
  Intubation PaFi<150 plus vasopressors or ECMO or Dialysis (9) | 0 | 0
  Intubation PaFi<150 or vasopressors (8) | 0 | 0
  Intubation PaFi<150 (7) | 0 | 1
  Hospitalized, NIV or high flow (6) | 0 | 0
  Hospitalized, mask or nasal prongs (5) | 1 | 0
  Hospitalized, no oxigen therapy (4) | 2 | 0
  Symptomatic, assistance needed (3) | 0 | 3
  Symptomatic, indeoendent (2) | 12 | 14
  Asymptomatic (1) | 42 | 38

ADVERSE EVENTS:
Time Frame: 90 days
Arm/Group | BOLUS | RECOVERY
All-Cause Mortality (participants affected / at risk) | 6/63 | 4/62
Serious Adverse Events (participants affected / at risk) | 22/63 | 21/62
Other Adverse Events (participants affected / at risk) | 25/63 | 15/62
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BOLUS (N=63) | RECOVERY (N=62)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 7 (7)
Hypertension (Cardiac disorders) | 1 (1) | 0 (0)
COVID worsering (Infections and infestations) | 9 (9) | 9 (9)
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
Pneumonia (Infections and infestations) | 6 (6) | 4 (4)
Sepsis (Infections and infestations) | 2 (2) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Thromboembolism (Vascular disorders) | 1 (1) | 3 (3) — Pulmonary thromboembolism
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BOLUS (N=63) | RECOVERY (N=62)
Hyperglycaemia (Endocrine disorders) | 15 (15) | 6 (6)
Rash (Immune system disorders) | 1 (1) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 1 (1)
Hypertension (Cardiac disorders) | 2 (2) | 1 (1)
Heart failure (Cardiac disorders) | 1 (1) | 1 (1)
Psychological/psychiatric disorders (Psychiatric disorders) | 3 (3) | 1 (1) — depressive anxiety disorder, confusion, depression...
Thrombotic disorders (Vascular disorders) | 1 (1) | 2 (2)
Tracheo-bronchitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Respiratory function worsering (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
* The sample size was not achieved due to the early termination of the study because of pandemia evolution.
* The open-label design and investigator-reported data on adverse events and infections may have led to bias in the description of these events.
* There was an imbalance in vaccination status between randomized groups.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-12-11): https://cdn.clinicaltrials.gov/large-docs/81/NCT04780581/Prot_SAP_000.pdf
  • Informed Consent Form (2021-01-07): https://cdn.clinicaltrials.gov/large-docs/81/NCT04780581/ICF_001.pdf